CLINICAL TRIAL: NCT01498497
Title: Six Month Safety Follow-up Study for PR-021 [Multicenter, Randomized, Double-blind, Placebo-controlled, Safety and Tolerability Phase 1/2a Study of Two Dosing Regimens of EUR-1100 for Oral Use, in Eosinophilic Esophagitis Subjects]
Brief Title: A Six Month, Safety Follow-up Study in Eosinophilic Esophagitis Subjects Who Completed Study PR-021
Status: Completed | Type: Observational
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-022
Record Dates: First submitted 2011-12-16; First posted 2011-12-23 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PR-021 Eosinophilic Esophagitis (EoE) Subjects: Subjects who received study drug and completed PR-021 study
  Interventions: Drug: EUR-1100; Drug: Placebo

INTERVENTIONS:
Drug: EUR-1100
Drug: Placebo

SUMMARY:
This purpose of this study is the long-term follow-up of glucocorticosteroid-related adverse events and hypothalamic-pituitary-adrenal axis (HPA) suppression in subjects after discontinuation of study drug received in the PR-021 study (Safety and Tolerability Study of Oral EUR-1100 to Treat Eosinophilic Esophagitis). The study will also provide the opportunity to better understand the natural course of eosinophilic esophagitis and define the treatment modalities of eosinophilic esophagitis with EUR-1100, such as the need for chronic maintenance or intermittent treatment.

All subjects who complete PR-021 will be offered the opportunity to participate in this study. The duration of this follow-up study is six months, during which subjects will visit the clinic for safety evaluation and clinical symptom assessment at the screening, Week 8, Week 16, and Week 24 visits. Additional phone visits will occur at Week 4, Week 12, and Week 20.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed full participation in Study PR-021 (Subjects discontinued prematurely from PR-021 due to HPA axis suppression will be eligible for study PR-022)
* Written informed consent (parent or legal guardian must sign when applicable) and assent form, if required
* Willing and able to adhere to all study procedures

Exclusion Criteria:

* Subjects already requiring medications or procedures for the treatment of EoE at the time of enrollment into the follow-up study, such as systemic (oral or parenteral) or inhaled corticosteroids, esophageal dilation, Proton Pump Inhibitors (PPIs) and/or dietary restrictions; in the case of subjects already on PPIs and /or dietary restrictions during Study PR-021, only subjects requiring an increase in dosage of PPIs and/or new dietary restrictions because of worsening of symptoms will be excluded
* Any physical, mental, or social condition, history or concurrent illness or laboratory abnormality that, in the investigator's judgment, might interfere with study procedures or the ability of the subject to adhere to and complete the study
* Contraindication to esophagogastroduodenoscopy (EGD) or esophageal biopsy or narrowing of the esophagus precluding EGD
* Female subjects who are pregnant or breastfeeding
* Participation in a clinical study involving an investigational drug or investigational device

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who received study drug and completed the PR-021 study (Safety and Tolerability Study of Oral EUR-1100 to Treat Eosinophilic Esophagitis)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Morning serum cortisol (change from baseline measure) | Baseline, Week 8, Week 16, and Week 24
Standard safety laboratory tests (change from baseline measure) | Baseline, Week 8, Week 16, and Week 24
  Hematology, serum chemistry, liver function tests, urinalysis, urine chemistry
Treatment-emergent adverse events collection (change from baseline measure) | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Physical examination and vital signs collection (change from baseline measure) | Baseline, Week 8, Week 16, and Week 24

SECONDARY OUTCOMES:
Esophagoduodenoscopy with multiple biopsies | Week 24
Patient reported outcomes and physician global assessment | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Ikuo Hirano, MD, Principal Investigator — Northwestern University School of Medicine
Locations (6):
- United States (6):
  - Children's Center for Digestive Health, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - South Jersey Pediatric Gastroenterology, Mays Landing, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania